CLINICAL TRIAL: NCT03877354
Title: Comparison of Tidal Volume Between Pediatric Anaesthesia and Paediatric Intensive Care Patients: Retrospective Study
Brief Title: Comparison of Tidal Volume Between Pediatric Anaesthesia and Paediatric Intensive Care Patients
Acronym: TIVAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2019/3
Record Dates: First submitted 2019-03-09; First posted 2019-03-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Protective Ventilation
Keywords: ventilation; paediatric patient; mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric patients anaesthesia: Paediatric patients who underwent diagnostic or surgical procedure under general anaesthesia with the need for mechanical ventilation in the selected time period.
  Interventions: Other: Data from anaesthesia records for ventilation setting screening
- Paediatric patients intensive care: Paediatric patients admitted to the paediatric intensive care unit with the need for mechanical ventilation in the selected time period
  Interventions: Other: Data from intensive care records for ventilation setting screening

INTERVENTIONS:
Other: Data from anaesthesia records for ventilation setting screening — Data from anaesthesia records will be retrospectively screened for the ventilation settings
  Other Names: Retrospective data analysis
  Groups: Paediatric patients anaesthesia
Other: Data from intensive care records for ventilation setting screening — Data from paediatric intensive care charts will be retrospectively screened for the ventilation settings
  Other Names: Retrospective data analysis
  Groups: Paediatric patients intensive care

SUMMARY:
Paediatric anaesthesiology and paediatric intensive care unit data will be retrospectively screened for the data regarding mechanical ventilation. The primary aim will be the tidal volume setting and the secondary the level of positive end-expiration pressure (PEEP) according to the inspired oxygen fraction (FIO2), and the level of driving pressure.

DETAILED DESCRIPTION:
Protective positive pressure ventilation (tidal volume ≤6 mL/kg) in adult patients in intensive care is currently considered as a standard procedure. It is associated with a reduction of morbidity and positive outcome. In paediatric patients there are available only limited information related to the size of the tidal volume and it is recommended to use the volume between 5 and 8 mL per kg for the whole spectrum of ages of pediatric patients. The aim of this retrospective observational study is to evaluate the tidal volumes used in clinical practice in pediatric patients during general anesthesia and compared it to the tidal volumes used in paediatric critical care. Data will be harvested from the anaesthesiology records and from the paediatric intensive care unit charts. The tidal volume will calculated per kg of actual weight.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients on mechanical ventilation in anaesthesia department
* Paediatric patients on mechanical ventilation in intensive care department
* In selected study period between 1.1.2018 - 31.1.2019

Exclusion Criteria:

* Age outside selected limits
* Insufficient data

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients on mechanical ventilation in anaesthesia departmentand in intensive care department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tidal volume | Intraoperative period
  Tidal volume will be evaluated in the paediatric patients in anaesthesia and in intensive care unit

SECONDARY OUTCOMES:
Positive end-expiratory pressure settings according to the inspiration fraction of oxygen | Intraoperative period
  Positive end-expiratory pressure will be evaluated in the paediatric patients in anaesthesia and in intensive care unit
Driving pressure | Intraoperative period
  Driving pressure will be calculated from peak pressure minus PEEP in patients on mechanical ventilation in anaesthesia and in intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, assoc.Prof.MD.Ph.D, Study Chair — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, State, Czechia

IPD SHARING:
Plan to Share IPD: Undecided